CLINICAL TRIAL: NCT03339960
Title: Ergonomics of Laparoscopy: Robotic Camera Controlled Versus Human Camera Controlled - A Randomized Controlled Trial
Brief Title: Ergonomics of Laparoscopy: Robotic Camera Controlled Versus Human Camera Controlled
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meander Medical Center (Other)
Collaborators: Wilhemina Ziekenhuis Assen (Unknown)
Responsible Party: Principal Investigator, Paul Wijsman, Study coordinator, Meander Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL61977.100.17
Record Dates: First submitted 2017-11-07; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic camera controlled (Active Comparator)
  Interventions: Other: Ergonomic measurement
- Human camera controlled (Active Comparator)
  Interventions: Other: Ergonomic measurement

INTERVENTIONS:
Other: Ergonomic measurement — Ergonomic measurement of the surgeon and assistant

SUMMARY:
Minimal invasive surgery has acquired increased importance and the number of procedures performed is ever growing. Laparoscopic surgery has several distinct key benefits for patients over open surgery and therefore it is considered as standard treatment for most general surgery procedures. These benefits include faster recovery, shorter hospital stay, reduced post-operative pain and improved cosmetic results.

However, laparoscopy has an increased burden to surgeons and many surgeons experience fatigue and physical discomforts due to laparoscopy. Robotic systems have been developed to improve the ergonomics (among other things), with good results. Many of the laparoscopy disadvantages have been overcome by robotic assisted surgery, such as increased range of motion, correction of the inverted instruments, and elimination of tremors.(4) Moreover, visualization of the operation is improved by personal camera control and stabilization of the image.

The AutoLap system, a video analytic robotic camera holder, has been developed to hold the camera in a stable manner. It enables the surgeon to control the camera and eliminates the need for coordination and communication between surgeon and assistants.

This study aims to evaluate the ergonomics of the surgeon and assistant during laparoscopy with the aid of the AutoLap system and compare it to standard laparoscopy. Also, it will be assessed whether the AutoLap can reduce physical and mental discomfort of both the surgeon and the assistant.

Objective This multicenter randomized controlled trial aims to compare ergonomics of the OR nurse and the surgeon during standard laparoscopic procedures with laparoscopic procedures aided by a robotic camera holder, the AutoLap system.

Study design Prospective, interventional, open, multicenter randomized controlled trial. The study will be conducted in Wilhemina Hospital Assen and in Meander Medical Center Amersfoort.

Study population

Adults ≥18 years who are scheduled for the following procedures:

* Laparoscopic hiatal hernia repair / fundoplication
* Laparoscopic right hemicolectomy
* Laparoscopic sigmoid resection
* Laparoscopic rectopexy
* Laparoscopic low anterior resection
* Laparoscopic splenectomy

Inclusion criteria

1. Aged ≥ 18 years
2. Fit for standard laparoscopic general surgery

Exclusion criteria

1. Contra-indications for laparoscopy
2. Obesity (BMI >35 Kg/m2)

Intervention AutoLap group: In the AutoLap group, the camera will be held by a robotic arm. Posture of the surgeon and the assistant will be recorded during standardized predefined steps of the procedure.

Control group: In the control group the camera will be held and maneuvered by a human assistant. The procedures will be performed according to the hospital and OR routine procedure. The surgical team will consist of 2 assistants and a surgeon. One of the assistants (OR-nurse, intern or resident) will hold the laparoscope and maneuver it. Posture of the surgeon and the assistant that maneuvers the laparoscope will be recorded during standardized predefined steps of the procedure.

Main study parameters/endpoints:

- RULA score, measured during predefined steps of the procedures.

Secondary parameters/endpoints:

- Questionnaires: Subjective Mental Effort Questionnaire (SMEQ), Local Experienced Discomfort (LED) scale (before and after the operation), NASA Task Load Index (NASA TLX).

DETAILED DESCRIPTION:
Objective:

It is our hypothesis that the ergonomics of the surgeon and his/her assistant will be improved with the aid of the AutoLap than without the aid of a robotic camera holder. Maintaining the same posture for a long period of time can lead to discomfort and fatigue of the surgeon and his/her assistant. Also, the space at the OR table is limited. Therefore, their body postures are sometimes awkward, unnatural and out of neutral position. With the aid of a robotic camera holder, we expect to minify this problem and improve ergonomics during laparoscopic operations.

The Autolap system is CE mark approved and is used frequently during laparoscopic operations. No patient characteristics and data will be recorded. The ethics committee MEC-U in Nieuwegein assessed this study and concluded that it does not fall under the scope of the WMO. Therefore this is non-WMO research.

The system shall be used in accordance with its cleared indication according to the clinical plan by clinical staff that has appropriate qualifications and training.

Predefined steps of the procedures:

The defined steps for a hiatal hernia repair / fundoplication are as follows:

* Opening of pars flaccida
* Deperitonialisation of the crura
* Resection of the hernia sac
* Suturing of the crura
* Dissection of the vasa brevia (if applicable)
* Creation of the fundoplication

The defined steps for a right hemicolectomy are as follows:

* Mobilisation of the coecum
* Dissection Toldt's line (lateral mobilization)
* Making the Subcolic tunnel
* Dissection of the ileo-colic artery
* Dissection of gastrocolic ligament
* Mobilization of the transverse colon
* Making the anastomosis (if performed laparoscopically)

The defined steps for a sigmoid resection are as follows:

* Dissection Toldt's line (lateral mobilization)
* Exposing the ureter
* Colon descendens mobilisation
* Mobilisation of flexura lienalis
* Dissecting the mesocolon
* Making the anastomosis (if performed laparoscopically)

The defined steps for a rectopexy are as follows:

* Incision of peritoneum over the promotorium
* Posterior resection behind the rectum
* Dissection towards pelvic floor
* Anterior resection of peritoneum
* Fixation of the mesh
* Removal of excess mesh
* Closing the peritoneum

The defined steps for a splenectomy are as follows:

* Opening of lesser peritoneal sac
* Division of gastrosplenic ligament
* Division of splenocolic ligament
* Division of pancreaticosplenic ligament
* Division of the hilum (vein and artery)
* Posterior and lateral dissection

The defined steps for a low anterior resection are as follows:

* Mobilisation of the sigmoid
* Dissection of the inferior mesenteric vena and arteria
* Dissection of the posterior wall of the mesorectum
* Lateral dissection of the sigmoid / rectum (freeing left colonic gutter)
* Dissection of the anterior wall of the rectum
* Dissection of Waldeyer's fascia
* Division of the distal rectum

Position and angles of the posture will be measured with MATLAB software. The posture of the surgeon and assistant will be photographed during the operation in two directions; from the side and from behind. These photographs will be used to calculate the RULA score. The RULA score is only measured during laparoscopic parts of the operation; if a part of the operation is performed open (not laparoscopically) RULA score will NOT be measured during the open part. No patient data or measurements will be acquired during this study. The positioning of the surgeon and operating assistant, operating table and OR monitors will be standardized for each type of procedure. Also, the placement of the monitors will be taken into account in such a way that a good ergonomic posture of the surgeon and assistant is ensured.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged ≥ 18 years
* 2) Fit for standard laparoscopic general surgery

Exclusion Criteria:

* 1) Contra-indications for laparoscopy
* 2) Obesity (BMI >35 Kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Mean Rapid Upper Limb Assessment score | Measured during predefined steps of the procedures
  Range: 1-7

SECONDARY OUTCOMES:
Mean Subjective Mental Effort Questionnaire | Directly after the surgery
  Range: 0-150
Mean Local Experienced Discomfort scale | Before and directly after the surgery
  Range: 0-10 per body part
Mean NASA Task Load Index | Directly after the surgery
  Range: 1-21 per dimension (7 in total)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Meander Medical Center, Amersfoort
  - Wilhemina Ziekenhuis Assen, Assen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijsman PJM, Molenaar L, Van't Hullenaar CDP, van Vugt BST, Bleeker WA, Draaisma WA, Broeders IAMJ. Ergonomics in handheld and robot-assisted camera control: a randomized controlled trial. Surg Endosc. 2019 Dec;33(12):3919-3925. doi: 10.1007/s00464-019-06678-1. Epub 2019 Feb 11. PMID 30746574